CLINICAL TRIAL: NCT04866381
Title: An Exploratory Clinical Study of SHR6390 and SHR1020 in the Treatment of Esophageal Squamous Cell Carcinoma After Progression on PD-1 Antibody
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIH-PQS-20210408
Record Dates: First submitted 2021-04-15; First posted 2021-04-29 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Esophageal Squamous Cell Carcinoma; Progression to PD-1 Antibody
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; famitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SHR-6390 (Experimental): SHR-6390
  Interventions: Drug: SHR-6390
- SHR-6390 combined with Camrelizumab (SHR-1210) (Experimental): SHR-6390 combined with Camrelizumab (SHR-1210)
  Interventions: Drug: SHR-6390 + Camrelizumab (SHR-1210)
- Camrelizumab (SHR-1210) combined with SHR-1020 (Experimental): Camrelizumab (SHR-1210) combined with SHR-1020
  Interventions: Drug: Camrelizumab (SHR-1210) + SHR-1020

INTERVENTIONS:
Drug: SHR-6390 — SHR-6390
  Arms: SHR-6390
Drug: SHR-6390 + Camrelizumab (SHR-1210) — SHR-6390 combined with Camrelizumab (SHR-1210)
  Arms: SHR-6390 combined with Camrelizumab (SHR-1210)
Drug: Camrelizumab (SHR-1210) + SHR-1020 — Camrelizumab (SHR-1210) combined with SHR-1020
  Arms: Camrelizumab (SHR-1210) combined with SHR-1020

SUMMARY:
This study is being conducted to explore the efficacy of SHR-6390 and SHR-1020 in the treatment of esophageal squamous cell carcinoma after progression on PD-1 Antibody.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed as esophageal squamous cell carcinoma by histopathology with at least one measurable lesion according to RECIST 1.1 criteria.
* Must have had progressive disease after previous treatment with PD-1 inhibitor
* ECOG score 0-2
* The expected survival time is ≥ 12 weeks
* Previous permanent discontinuation did not occur due to adverse events associated with immunotherapy, or the immunotreatment-related adverse events recovered to ≤1 grade

Exclusion Criteria:

* Had other active malignant tumors within 5 years before entering the study
* Had abnormal swallowing function or dysfunction of gastrointestinal absorption
* The first study drug treatment was less than 28 days or 5 half-lives (in terms of longer) from the last radiotherapy, chemotherapy, targeted therapy or immunotherapy
* Patients who have already received surgery within 28 days (biopsy for diagnosis is permitted)
* Pregnant or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 1 year
  Objective Response Rate is defined as the percentage of patients whose tumors have a complete or partial response to treatment among eligible and treated patients. Objective response rate is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1 criteria.

SECONDARY OUTCOMES:
Progression-Free-Survival | Up to 1 year
  Progression-Free-Survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first.
Overall survival | Up to 1 year
  Overall survival is defined as time from treatment start date to date of death from any cause. Patients alive at the time of analysis are censored at last contact date.
Subject safety | Up to 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No